CLINICAL TRIAL: NCT03490734
Title: Neurobehavioral Plasticity to Regular Sugar-Sweetened Beverage Intake: An fMRI Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17-0710; 1R01DK112317-01A1 (NIH)
Record Dates: First submitted 2018-03-15; First posted 2018-04-06 (Actual); Results first posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Weight Gain
Keywords: nutrition; obesity; weight gain; sugar; sugar sweetened beverage; dopamine; neurobehavioral adaptation
MeSH Terms: conditions — Obesity; Weight Gain | interventions — Water

STUDY DESIGN:
Intervention Model Description: Stratified randomization techniques will be used to distribute: 1) male & females, 2) those with a BMI > 26.1 & those with a BMI < 26.1, and 3) regular SSB consumers (> 1/day; 12 fl oz) & low or non-SSB consumers equally across the 2 experimental conditions (SSB vs. unsweetened beverage) and then to the two flavors within each experimental condition. BMI of 26.0 was selected as it is the midpoint of inclusion criteria 18 < BMI < 34.
Who Masked: Participant
Masking Description: Experimental and flavor conditions will be blinded to those performing analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Beverage A (Sweetened) (Active Comparator): One quarter of the group to receive black cherry and orange flavored beverage with added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a water solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Interventions: Dietary Supplement: Black Cherry and Orange Flavored Beverage with added sugar; Other: Water
- Beverage B (Sweetened) (Active Comparator): One quarter of the group to receive strawberry kiwi & lemonade flavored beverage with added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a water solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Interventions: Dietary Supplement: Strawberry Kiwi &Lemonade Flavored Beverage with added sugar; Other: Water
- Beverage A (Unsweetened) (Active Comparator): One quarter of the group to receive black cherry and orange flavored beverage no added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a water solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Interventions: Dietary Supplement: Black Cherry and Orange Flavored Beverage no added sugar; Other: Water
- Beverage B (Unsweetened) (Active Comparator): One quarter of the group to receive strawberry kiwi & lemonade flavored beverage no added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a water solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Interventions: Dietary Supplement: Strawberry Kiwi & Lemonade Flavored Beverage no added sugar; Other: Water

INTERVENTIONS:
Dietary Supplement: Black Cherry and Orange Flavored Beverage with added sugar — 10 oz daily for three weeks
  Other Names: Kool-Aid®
  Arms: Beverage A (Sweetened)
Dietary Supplement: Strawberry Kiwi &Lemonade Flavored Beverage with added sugar — 10 oz daily for three weeks
  Other Names: Kool-Aid®
  Arms: Beverage B (Sweetened)
Dietary Supplement: Black Cherry and Orange Flavored Beverage no added sugar — 10 oz daily for three weeks
  Other Names: Kool-Aid®
  Arms: Beverage A (Unsweetened)
Dietary Supplement: Strawberry Kiwi & Lemonade Flavored Beverage no added sugar — 10 oz daily for three weeks
  Other Names: Kool-Aid®
  Arms: Beverage B (Unsweetened)
Other: Water — Three mL administered per associated logo presentation only during MRI procedure.

SUMMARY:
The proposed project will examine the strength, specificity and persistence of neurobehavioral adaptions that occur in the initial period of repeated consumption of a branded sugar sweetened beverage (SSB).

DETAILED DESCRIPTION:
The proposed project addresses critical gaps in the understanding of the strength, specificity and persistence of neurobehavioral adaptions that occur in the initial period of repeated consumption of a branded sugar sweetened beverage (SSB). Half of Americans consume SSBs on any given day.

Regular SSB intake is considered a contributing factor to excess energy intake, weight gain, and obesity, which impacts 70% of Americans. A contributing factor to repeated SSB consumption is sugar intake causes the release of dopamine (DA) and opioids in the striatum, providing positive reinforcement. As such, multiple brain-based models of food reward-driven obesity have been proposed, largely focusing on the striatum and executive functioning. These brain-based models of obesity have elucidated risk factors for overconsumption of high-sugar foods; however, data supporting these competing models rely heavily on observational studies in small samples.

Importantly, previous reports from the investigators lab and others directly implicate eating behavior patterns as a vital contributor to aberrant neurobehavioral responses to food stimuli. However, without experimental evidence, there are fundamental gaps in the investigators knowledge about the neurobehavioral adaptations that occur as an individual begins to regularly consume a SSB prior to weight change.

As observational data suggest, it is also crucial to examine individual difference factors that may exacerbate or protect against adaptations associated with regular SSB intake, as well as whether these adaptions are specific.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants will be eligible for the study if they have BMI scores between the 18 and 34 at baseline.

Exclusion Criteria:

* Individuals with probable current Axis I psychopathology or any fMRI contra-indicators (e.g., metal implants, braces) will be excluded. Those with a probable Axis I diagnosis will be provided with treatment referral information and encouraged to seek treatment,
* current regular use (3 or more times a week) of psychoactive drugs (e.g., cocaine, marijuana, nicotine),
* regular smoking,
* serious medical problems (e.g., cancer, diabetes),
* dietary practices that do not allow intake of intervention beverages.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Burger, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Mcgavran-Greenberg Hall, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Peirce JW. PsychoPy--Psychophysics software in Python. J Neurosci Methods. 2007 May 15;162(1-2):8-13. doi: 10.1016/j.jneumeth.2006.11.017. Epub 2007 Jan 23. PMID 17254636

RESULTS

PARTICIPANT FLOW:
Groups:
- Beverage A (Sweetened): One quarter of the group to receive black cherry and orange flavored beverage with added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a water solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Black Cherry and Orange Flavored Beverage with added sugar: 10 oz daily for three weeks
  Water Solution: Three mL administered per associated logo presentation only during MRI procedure.
- Beverage B (Sweetened): One quarter of the group to receive strawberry kiwi & lemonade flavored beverage with added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a water solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Strawberry Kiwi &Lemonade Flavored Beverage with added sugar: 10 oz daily for three weeks
  Water Solution: Three mL administered per associated logo presentation only during MRI procedure.
- Beverage A (Unsweetened): One quarter of the group to receive black cherry and orange flavored beverage no added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a water solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Black Cherry and Orange Flavored Beverage no added sugar: 10 oz daily for three weeks
  Water Solution: Three mL administered per associated logo presentation only during MRI procedure.
- Beverage B (Unsweetened): One quarter of the group to receive strawberry kiwi & lemonade flavored beverage no added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a water solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Strawberry Kiwi & Lemonade Flavored Beverage no added sugar: 10 oz daily for three weeks
  Water Solution: Three mL administered per associated logo presentation only during MRI procedure.
Period: Pre-intervention Baseline Visit
Arm/Group | Beverage A (Sweetened) | Beverage B (Sweetened) | Beverage A (Unsweetened) | Beverage B (Unsweetened)
Started | 47 | 38 | 34 | 41
Completed | 47 | 38 | 34 | 41
Not Completed | 0 | 0 | 0 | 0
Period: Pre-intervention Scan Visit
Arm/Group | Beverage A (Sweetened) | Beverage B (Sweetened) | Beverage A (Unsweetened) | Beverage B (Unsweetened)
Started | 47 | 38 | 34 | 41
Completed | 45 | 37 | 34 | 37
Not Completed | 2 | 1 | 0 | 4
Not completed — fMRI contraindications | 2 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Post-intervention Scan Visit
Arm/Group | Beverage A (Sweetened) | Beverage B (Sweetened) | Beverage A (Unsweetened) | Beverage B (Unsweetened)
Started | 45 | 37 | 34 | 37
Completed | 43 | 34 | 34 | 34
Not Completed | 2 | 3 | 0 | 3
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 3
Period: Post-intervention Behavioral Visit
Arm/Group | Beverage A (Sweetened) | Beverage B (Sweetened) | Beverage A (Unsweetened) | Beverage B (Unsweetened)
Started | 43 | 34 | 34 | 34
Completed | 43 | 34 | 34 | 34
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Beverage A (Sweetened) | Beverage B (Sweetened) | Beverage A (Unsweetened) | Beverage B (Unsweetened) | Total
Number analyzed (Participants) | 47 | 38 | 34 | 41 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.9 (2.5) | 21.4 (2.3) | 21.9 (2.4) | 21.3 (2.5) | 21.6 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 22 | 21 | 24 | 96
  Male | 18 | 16 | 13 | 17 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 5 | 2 | 17
  Not Hispanic or Latino | 42 | 33 | 29 | 39 | 143
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 12 | 5 | 7 | 15 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 2 | 1 | 13
  White | 25 | 24 | 22 | 22 | 93
  More than one race | 3 | 2 | 0 | 1 | 6
  Unknown or Not Reported | 2 | 2 | 3 | 2 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 38 | 34 | 41 | 160
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.4 (3.5) | 23.1 (2.7) | 23.9 (3.5) | 22.7 (3.0) | 23.2 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Voxel-wise Blood Oxygen Level Dependent (BOLD) Including Outliers Using Functional Magnetic Resonance Imaging (fMRI) of Brain Activation Signals in Response to Beverage Taste and Logo
Description: The fMRI paradigm assesses evoked blood oxygen level dependent (BOLD) response to receipt of study beverages (sweet and unsweet) and a water solution, and logo-elicited anticipation of both beverages and water solution. The visual stimuli are two beverage logos, a water logo, and a fixation cross. Each logo (1 second) signals impending delivery of 3 mL of the associated juice/water over 6 seconds, with the fixation cross otherwise presented. A jitter ranging from 5 to 13 seconds follows each trial. In total, the participants are shown 24 repeats of the events of interest over 4, 7-minute runs. Contrasts of interest are the post- > pre-intervention BOLD response to sweetened beverage logo > water logo. Parameter estimates for these contrasts are extracted and reported. A positive reported outcome reflects higher post- vs. pre-intervention (negative values reflect lower post- vs. pre-intervention) change in whole-brain BOLD response for sweetened beverage logo > water logo for each arm.
Time Frame: Baseline and Post-intervention Assessment. Post-Intervention Assessment completed approximately 5 weeks after the Baseline Assessment
Population: Decrease in the sample was due to missing data and/or errors in neuroimaging data processing.
  For results reporting, the two types of flavored beverages (strawberry, kiwi & lemonade OR black cherry & orange) were combined based on sweetness (sweetened vs. unsweetened beverage) resulting in two arms. We combined beverages across flavors, since the main outcome of interest is the effect of sugar in beverages independent of flavor.
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- Beverages A (Sweetened) and B (Sweetened): Half of the group to receive a flavored beverage (strawberry, kiwi & lemonade flavored OR black cherry & orange flavored) with added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a water solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Black Cherry and Orange Flavored Beverage with added sugar: 10 oz daily for three weeks OR Strawberry Kiwi &Lemonade Flavored Beverage with added sugar: 10 oz daily for three weeks
  Water Solution: Three mL administered per associated logo presentation only during MRI procedure.
- Beverages A (Unsweetened) and B (Unsweetened): Half of the group to receive a flavored beverage (strawberry, kiwi & lemonade flavored OR black cherry & orange flavored) no added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a water solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Black Cherry and Orange Flavored Beverage no added sugar: 10 oz daily for three weeks OR Strawberry Kiwi &Lemonade Flavored Beverage no added sugar: 10 oz daily for three weeks
  Water Solution: Three mL administered per associated logo presentation only during MRI procedure.
Arm/Group | Beverages A (Sweetened) and B (Sweetened) | Beverages A (Unsweetened) and B (Unsweetened)
Number analyzed (Participants) | 64 | 58
arbitrary units | -2.69 (13.52) | -3.06 (14.89)
Statistical Analysis 1: Comparison: Beverages A (Sweetened) and B (Sweetened) vs Beverages A (Unsweetened) and B (Unsweetened); Whole-brain analyses were used. No clusters of significant activation were detected; Test type: Superiority; p = 0.52, ANCOVA — Corrected for multiple comparisons by using the threshold free cluster enhancement, nonparametric thresholding algorithm in FMRIB Software Library (FSL), resulting in a family-wise error rate (FWE) corrected significance threshold of p-FWE<0.05

2. Secondary Outcome: Change in Voxel-wise Blood Oxygen Level-Dependent (BOLD) Brain Activation in Response to Beverage Taste and Logo by Body Mass Index (BMI)
Description: The fMRI paradigm assesses evoked blood oxygen level dependent (BOLD) response to receipt of study beverages, (sweetened and unsweetened) and a water solution, and logo-elicited anticipation of both beverages and water solution. Whole-brain analyses are performed. Contrasts of interest for the within-subject models are post-intervention > pre-intervention BOLD response to beverage vs. water logo and contrasts of interest for the group model are sweetened beverage logo > water logo. To test the interaction of brain activation with BMI, BMI is entered as a covariate in the group model. Parameter estimates of significant BOLD response to these contrasts are extracted and reported. A positive reported outcome reflects higher post- vs. pre-intervention (negative values reflect lower post- vs. pre-intervention) change in BOLD response in the putamen for the sweetened beverage logo > water logo for each arm.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Beverages A (Sweetened) and B (Sweetened) | Beverages A (Unsweetened) and B (Unsweetened)
Number analyzed (Participants) | 64 | 58
arbitrary units | 3.47 (204.99) | -9.82 (198.96)
Statistical Analysis 1: Comparison: Beverages A (Sweetened) and B (Sweetened) vs Beverages A (Unsweetened) and B (Unsweetened); Test type: Superiority; p = 0.016, ANCOVA — Corrected for multiple comparisons by using the threshold free cluster enhancement (TFCE), nonparametric thresholding algorithm in FSL, resulting in a family-wise error rate corrected significance threshold of p-FWE < 0.05

3. Secondary Outcome: Beverage Perceptual Ratings Using Visual Analog Scales
Description: Perceptual ratings of the assigned beverage using visual analog scales are assessed at the pre- and post-intervention behavioral visits.
  Visual analog scales (VAS) are presented on an iPad screen. The scale assesses response to taste after the participant consumes a small amount of the beverage. Perceived pleasantness of, and desire to consume the two beverages is measured using adapted labeled hedonic scales at pre-/post-intervention. Pleasantness is phrased 'How pleasant is this taste' and anchored by (-100) 'most unpleasant imaginable' to (100) 'most pleasant imaginable', and 'neutral' (0) in the middle. Desire follows a similar pattern using 'desire to consume' as the phrasing. Pleasantness and desire of the assigned beverage is also evaluated at the 9 intervention assessments. Higher scores represent higher pleasantness and desire.
Time Frame: Pre-intervention Behavioral Assessment; Post-intervention Behavioral Assessment; Post-intervention Assessment completed approximately 5 weeks after the Pre-intervention Assessment
Population: Decrease in the sample was due to missing data.
  For results reporting, the two types of flavored beverages (strawberry, kiwi & lemonade OR black cherry & orange) were combined based on sweetness (sweetened vs. unsweetened beverage) resulting in two arms. We combined beverages across flavors, since the main outcome of interest is the effect of sugar in beverages independent of flavor.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Beverages A (Unsweetened) & B (Unsweetened): Half of the group to receive a flavored beverage (strawberry, kiwi & lemonade flavored OR black cherry & orange flavored) no added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a water solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Black Cherry and Orange Flavored Beverage no added sugar: 10 oz daily for three weeks OR Strawberry Kiwi &Lemonade Flavored Beverage no added sugar: 10 oz daily for three weeks
  Water Solution: Three mL administered per associated logo presentation only during MRI procedure.
Arm/Group | Beverages A (Sweetened) and B (Sweetened) | Beverages A (Unsweetened) & B (Unsweetened)
Number analyzed (Participants) | 64 | 58
score on a scale
  Pre-Intervention "Pleasantness" ratings of assigned beverage | 25.00 (3.20) | -21.00 (3.30)
  Post-Intervention "Pleasantness" ratings of assigned beverage | 24.20 (3.60) | -8.84 (3.80)
  Pre-Intervention "Desire to consume" ratings of assigned beverage | 20.30 (3.50) | -23.70 (3.60)
  Post-Intervention "Desire to consume" ratings of assigned beverage | 22.90 (3.90) | -12.20 (4.10)

4. Secondary Outcome: Stop Signal Reaction Time to Logo as Measured by Behavioral Response Inhibition Task
Description: Stop-signal reaction time to assigned beverage logo are assessed at the pre- and post-intervention visits.
  The behavioral response inhibition task (stop-signal task) examines motor disinhibition in response to beverage logos. This allows for the assessment of bias toward the logos and is sensitive to detect changes due to the intervention. The task is performed on an iPad app where participants complete the task twice, once at the pre-intervention and once at the post-intervention behavioral visit. The task contains 6 runs, where 3 runs present the logo of the assigned beverage and the other 3 present the logo of the same-flavor unassigned beverage. Within each run of this task, 64 (20 "go") trials are presented, and participants are instructed to make a speeded response to a "go" stimulus except for trials when a "stop" signal occurs (an X presented over the logo), in which case participants are instructed to withhold their response.
Time Frame: as for outcome 3
Population: Missing data occurred due to errors with the stop-signal task on the ipad.
  For results reporting, the two types of flavored beverages (strawberry, kiwi & lemonade OR black cherry & orange) were combined based on sweetness (sweetened vs. unsweetened beverage) resulting in two arms. We combined beverages across flavors, since the main outcome of interest is the effect of sugar in beverages independent of flavor.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Beverages A (Sweetened) and B (Sweetened) | Beverages A (Unsweetened) and B (Unsweetened)
Number analyzed (Participants) | 48 | 39
seconds
  Pre-intervention reaction time | 0.5321 (0.0654) | 0.5452 (0.0850)
  Post-intervention reaction time | 0.5013 (0.0609) | 0.5360 (0.1057)

5. Other Pre Specified Outcome: Percent Change in Voxel-wise Blood Oxygen Level Dependent (BOLD) Including Outliers Using Functional Magnetic Resonance Imaging (fMRI) of Brain Activation Signals in During Rest
Description: The investigators use resting state fMRI (rsfMRI) data to assess intrinsic functional connectivity and network analyses. Functional connectivity is commonly quantified by measuring the synchronization of low-frequency BOLD fluctuations across pairs of brain regions of interest (ROIs) via correlation coefficients (see statistical analyses). rsfMRI data is acquired in one run of 7 minutes; participants are asked to remain still with their eyes open, and to fixate on the fixation cross.
Time Frame: Baseline Assessment; Post-Intervention Assessment, Post-Intervention Assessment completed approximately 5 weeks after the Baseline Assessment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Modulation of Blood Oxygen Level Dependent (BOLD) Using Functional Magnetic Resonance Imaging (fMRI) of Brain Activation Signals in Response to Beverage Taste and Logo by TaqIA Single Nucleotide Polymorphism Status
Description: Saliva from participants is used to extract DNA using standard salting-out and solvent precipitation methods, to yield an average of 45 µg of DNA. The TaqIA (rs1800497) assays are done using a fluorogenic 5_nuclease (Taqman, ABI) method on an ABI Prism 7000 Sequence Detection System via the allelic discrimination mode. Reactions containing 20ng of DNA are performed in 10 µl reactions with TaqMan Universal Polymerase Chain Reaction Master Mix using standard cycling conditions. Independent investigators score allele sizes; inconsistencies are reviewed and rerun when necessary. For every assay, each 96-well plate includes non-template and DNA standards of known genotype. All genotyping is performed at the UNC-CH Advanced Analytics Core
Time Frame: as for outcome 5
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Food Pattern From Baseline to Post-Intervention Assessment by Food Frequency Questionnaire
Description: The Food Frequency Questionnaire (FFQ) is a self-reported checklist of 76 foods and beverages with a frequency response section. Subjects report generally how often each item is consumed over a two-week period of time. The six possible responses are 1= never in the last two weeks, 2= 1-3 times in the last 2 weeks, 3= 4-6 times in the last 2 weeks, 4= 7-9 times in the last two weeks, 5= 10-13 times in the last 2 weeks, 6= daily or more in the last two weeks. Response information is used to estimate daily caloric intake (number of kcal) and macronutrient content (percent calories from carbohydrate/fat/protein). Food pattern is assessed as an aggregate of these measures. Changes in food pattern will be assessed as a difference from baseline to post-intervention assessment.
Time Frame: as for outcome 5
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Beverage Intake Pattern From Baseline to Post-Intervention Assessment by Beverage Intake Questionnaire
Description: To better capture variation in regular beverage intake patterns, the Beverage Intake Questionnaire is administered which queries directly about intake of all types of beverages. Similar to the Food Frequency Questionnaire, subjects report generally how often each item is consumed over a two-week period of time. The possible responses are 1= never in the last two weeks, 2= 1-3 times in the last 2 weeks, 3= 4-6 times in the last 2 weeks, 4= 7-9 times in the last two weeks, 5= 10-13 times in the last 2 weeks, 6= daily or more in the last two weeks. Responses information is used to estimate daily caloric intake from beverages (number of kcal) and macronutrient content (number of calories from carbohydrate/fat/protein). Changes in beverage intake are assessed as a difference from baseline to post-intervention assessment.
Time Frame: as for outcome 5
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Physical Activity From Baseline to Post-Intervention Assessment by the Short-Form International Physical Activity Questionnaire
Description: The International Physical Activity Questionnaire (IPAQ), which has shown high test-retest reliability, assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives and estimates total physical activity in metabolic equivalent of task (MET-min/week) and time spent sitting. Changes in physical activity are assessed as a difference from pre- to post-intervention assessment.
Time Frame: as for outcome 5
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Restrained Eating Subscale Score as Measured on Dutch Eating Behavior Questionnaire
Description: The Dutch Eating Behavior Questionnaire is a 33-item self-report measure designed to assess the type of eating behavior and is organized into 3 subscales (emotional eating, externally-induced eating, and restrained eating). Subjects rate the frequency of their eating behaviors using a 5-point scale, where 1=never, 2=seldom, 3=sometimes, 4=often, and 5=very often. The Restrained Eating subscale consisted of 10 items and the scores range from 10 (worse outcome) to 50 (better outcome). The change is calculated as the difference between scores at Baseline and Post-Intervention Assessment.
Time Frame: as for outcome 5
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Food Craving as Assessed by the Food Craving Inventory (FCI) Score Changes of Food Pattern From Baseline by Food Frequency Questionnaire During the Intervention
Description: The Food Craving Inventory is a 28-item instrument measuring the frequency over the past month of general cravings and cravings for specific types of foods, namely: high fats, sweets, carbohydrates/starches, and fast-food fats. Subjects rate how often they have experienced a craving for each food on a 5-point frequency scale, where 1=never, 2=rarely (once or twice), 3=sometimes, 4= often, 5= always/almost every day. Food craving score is calculated as a total sum, and the change score is calculated from the difference between baseline to post-intervention assessment.
Time Frame: as for outcome 5
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Hedonic Hunger as Assessed by the Power of Food Scale (PFS) Score
Description: The Power of Food scale assesses reported appetitive drive, food reward responsivity, sensitivity to food cues in the environment, and the frequency of food-related thoughts. The 21-item scale prompts subjects to rate how much they agree with statements about hedonic hunger on a 5-point scale, where 1=do not agree at all, 2=agree a little, 3=agree somewhat, 4=agree, and 5=strongly agree. The change in total PFS score will be calculated from the difference between baseline to post-intervention assessment.
Time Frame: as for outcome 5
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Food Habits as Assessed by the Yale Food Addiction Scale
Description: The Yale Food Addiction Scale (YFAS) is designed to identify participants who exhibit signs of possible food addiction to specific foods. The 9-item questionnaire is based on substance dependence criteria in the DSM-IV-TR, as well as on scales that are used to assess behavioral addictions. Subjects rate how often they have experienced a possible food addictive behavior on a 5-point frequency scale, where 0=never, 1=once a month, 2=2-4 times per month, 3= 2-3 times per week, 4= 4+ times per week. The change in total score is calculated from the difference between baseline to post-intervention assessment.
Time Frame: as for outcome 5
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in General Impulsivity as Assessed by the Barrett Impulsiveness Scale
Description: The Barratt Impulsiveness Scale is one of the most commonly used self-report measures of impulsivity. This instrument comprises 15 items that assess three independent sub-dimensions of impulsivity: (a) Attention; (b) Non-planning; (c) Motor. Collectively, the three sub-dimensions represent a total impulsivity score. Items are statements about behavior and participants rate each item are scored from 1 (Rarely/Never) to 4 (Almost Always/Always). The change in total score is calculated from the difference between baseline to post-intervention assessment.
Time Frame: as for outcome 5
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in General Sensitivity to Reward and Sensitivity to Punishment as Assessed by the Sensitivity to Punishment and Sensitivity to Reward Questionnaire
Description: The Sensitivity to Punishment/Sensitivity to Reward Questionnaire (SPSRQ) is a self-reported instrument that includes 48 yes/no questions divided into two subscales: Sensitivity to Reward (SR) and Sensitivity to Punishment (SP). Items statements about behavior, and participants will rate each item are scored from 1 (Definitely True) to 5 (Definitely False). The change in total score is calculated from the difference between baseline to post-intervention assessment.
Time Frame: as for outcome 5
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in Behavioral Approach and Behavioral Inhibition as Assessed by the BIS/BAS Scales
Description: The BIS/BAS scales are designed to assess individual differences in the sensitivity of two systems: A behavioral avoidance (or inhibition) system (BIS) and a behavioral approach system (BAS). The questionnaire includes 24 items. Items are statements about behavior and participants rate each item are scored from 1 (very true for me) to 4 (very false for me). The change in total score is calculated from the difference between baseline to post-intervention assessment.
Time Frame: as for outcome 5
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse data were collected for the duration (beginning to end) of each of the 4 study assessments (pre-intervention baseline visit, pre-intervention scan visit, post-intervention scan visit, post-intervention behavioral visit) and for the duration of the intervention (21 days), an average of 25 days.
Groups:
- Beverage A (Sweetened): One quarter of the group to receive black cherry and orange flavored beverage with added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a tasteless beverage solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Black Cherry and Orange Flavored Beverage with added sugar: 10 oz daily for three weeks
  Tasteless Beverage: A solution of water, potassium chloride, and sodium bicarbonate. Three mL administered per associated logo presentation only during MRI procedure.
- Beverage B (Sweetened): One quarter of the group to receive strawberry kiwi & lemonade flavored beverage with added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a tasteless beverage solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Strawberry Kiwi &Lemonade Flavored Beverage with added sugar: 10 oz daily for three weeks
  Tasteless Beverage: A solution of water, potassium chloride, and sodium bicarbonate. Three mL administered per associated logo presentation only during MRI procedure.
- Beverage A (Unsweetened): One quarter of the group to receive black cherry and orange flavored beverage no added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a tasteless beverage solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Black Cherry and Orange Flavored Beverage no added sugar: 10 oz daily for three weeks
  Tasteless Beverage: A solution of water, potassium chloride, and sodium bicarbonate. Three mL administered per associated logo presentation only during MRI procedure.
- Beverage B (Unsweetened): One quarter of the group to receive strawberry kiwi & lemonade flavored beverage no added sugar for 3 weeks.
  MRIs will be performed before starting and then after 3 weeks of daily beverage consumption wherein participants will be presented with visual stimuli of two beverage logos, one representing a tasteless beverage solution and another representing the assigned beverage. Each 1-second presentation signals impending delivery of 3 mL of the associated beverage via a plastic mouthpiece during MRI.
  Strawberry Kiwi & Lemonade Flavored Beverage no added sugar: 10 oz daily for three weeks
  Tasteless Beverage: A solution of water, potassium chloride, and sodium bicarbonate. Three mL administered per associated logo presentation only during MRI procedure.
Arm/Group | Beverage A (Sweetened) | Beverage B (Sweetened) | Beverage A (Unsweetened) | Beverage B (Unsweetened)
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/38 | 0/34 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/38 | 0/34 | 0/41
Other Adverse Events (participants affected / at risk) | 2/47 | 0/38 | 0/34 | 0/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Beverage A (Sweetened) (N=47) | Beverage B (Sweetened) (N=38) | Beverage A (Unsweetened) (N=34) | Beverage B (Unsweetened) (N=41)
nausea during fMRI scan (Gastrointestinal disorders) | 2 (2) | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT03490734/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT03490734/SAP_001.pdf